CLINICAL TRIAL: NCT00613470
Title: Pharmacodynamics and Pharmacokinetics of Citalopram and Escitalopram
Acronym: PGRN-SSRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Daniel K. Hall-Flavin, MD, Assistant Professor of Psychiatry, College of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 170-05; U01GM061388 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Depression
Keywords: Depression; Antidepressants
MeSH Terms: conditions — Depression | interventions — Citalopram; Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Citalopram and escitalopram (Experimental): Citalopram tablet or solution starting at 20 mg, increase to 40 mg at 4 weeks if QIDS-C16 > 5, keep at same dose if QIDS-C16 < 5.
  Escitalopram tablets starting at 10 mg, increase to 20 mg at 4 weeks if QIDS-C16 > 5, keep at same dose if QIDS-C16 < 5.
  Interventions: Drug: citalopram and escitalopram

INTERVENTIONS:
Drug: citalopram and escitalopram — escitalopram tablets starting at 10 mg, increase to 20 mg at 4 weeks if QIDS-C16 > 5, keep at same dose if QIDS-C16 < 5.
  citalopram tablet or solution starting at 2o mg, increase to 40 mg at 4 weeks if QIDS-C16 > 5, keep at same dose if QIDS-C16 < 5.

SUMMARY:
This study is one component of a larger U01 grant that was submitted in August, 2004 to the NIGMS as part of the Pharmacogenomic Research Network. This study will enroll 1200 patients over 4 years.

It is known that functionally significant genetic polymorphisms for the cytochrome P450 (CYPs) can contribute to individual differences in response to specific selective serotonin reuptake inhibitors (SSRIs). However, a better understanding of the pharmacogenomics of both PK and PD for SSRI antidepressants will inform clinical practice. Therefore, we propose to evaluate the contribution of pharmacogenomics to variation in response to the highly specific SSRIs citalopram (a racemic mixture) and escitalopram (a chiral compound containing the active S-isomer of citalopram ) by correlating both PK and PD variation for these agents with intragene haplotypes in genes encoding proteins involved in citalopram metabolism, as well as central nervous system (CNS) pathways for monoamine neurotransmitter biosynthesis, metabolism, storage, release, reuptake, and receptors. In the future this "candidate pathway" intragene haplotype genotyping strategy will also be complemented by the application of genome-wide screens performed with DNA from subjects with extreme phenotypes for response to citalopram.

Phenotypes to be measured before and after the initiation of citalopram or escitalopram therapy will include determinations of serum citalopram and metabolite concentrations, treatment response as measured by Hamilton Rating Scale for Depression indices, and number and severity of side effects as determined by structured questionnaires. The hypothesis to be tested is that inherited variation in citalopram metabolism and transport (PK) and/or PD variation as a result of inherited variation in monoamine neurotransmitter biosynthesis, metabolism, reuptake, storage, receptors or signaling contribute to individual variation in citalopram antidepressant efficacy and/or side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients or inpatients with nonpsychotic MDD.
2. A score of >14 on the HRS-D17 (equivalent to 10 or greater on PHQ-9 which is used in primary care to assess depression) given that when medication exceeds the effect of placebo in primary care participants have a HRS-D17 >12. We added 2 HRS-D17 points to take into account the possibility of measurement error.
3. Outpatients or inpatients for whom antidepressant treatment is deemed appropriate by the treating clinician.
4. Subjects who are between 18-85 years of age.
5. Participants who have general medical conditions (GMCs) which could conceivably be physiologically causing their depressive symptoms will receive treatment as usual for their GMCs as well as for their MDD.

Exclusion Criteria:

* Subjects with medical contraindications that preclude citalopram or escitalopram treatment and those who have previously failed to respond to citalopram or escitalopram will be excluded. In addition, patients with schizophrenia, schizoaffective disorder, or who have Bipolar I disorder will be excluded because they have a primary psychiatric condition that requires a different initial treatment. Subjects currently on antidepressant medication with subtherapeutic results in terms of depression management will undergo a medication taper and discontinuation prior to initiation of citalopram or escitalopram treatment. The subject will be closely monitored by the primary physician or psychiatrist during the medication taper and discontinuation phase. The medication taper is left upto the treating physician's or psychiatrist's discretion. Study subjects who cannot be safely tapered from their medication or experience adverse effects during the taper will be excluded from the study. Study subjects using their antidepressant medication for management of nicotine dependence, chronic pain, migraine prophylaxis or other diagnoses will not be eligible for the study. Trazodone, Melatonin, and Diphenhydramine may be used as rescue medications for insomnia. Benzodiazepines may be used for treatment of anxiety and atomoxetine may be used for the treatment of attention deficit disorder. Study subjects currently on antipsychotic medications (e.g., typical and atypical antipsychotic drugs) and mood stabilizing agents (e.g., lithium, carbamazepine, valproate, lamotrigine, gabapentin, or other anticonvulsants) are not eligible for the study with the exception of those starting quetiapine after baseline. Subjects unable to give informed consent are excluded. Pregnant subjects will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 927 (Actual)
Dates: Start 2005-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The change in HRS-D17 will constitute the major research outcome measure used to assess drug response phenotype because it is widely used in psychiatric research, making it possible to perform comparisons with other studies. | baseline, 4 week and 8 week visits

SECONDARY OUTCOMES:
QIDS-C16 (obtained by the CRC), and the QIDS-SR16 | week 0, 4, and 8

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K Hall-Flavin, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Liu D, Ray B, Neavin DR, Zhang J, Athreya AP, Biernacka JM, Bobo WV, Hall-Flavin DK, Skime MK, Zhu H, Jenkins GD, Batzler A, Kalari KR, Boakye-Agyeman F, Matson WR, Bhasin SS, Mushiroda T, Nakamura Y, Kubo M, Iyer RK, Wang L, Frye MA, Kaddurah-Daouk R, Weinshilboum RM. Beta-defensin 1, aryl hydrocarbon receptor and plasma kynurenine in major depressive disorder: metabolomics-informed genomics. Transl Psychiatry. 2018 Jan 10;8(1):10. doi: 10.1038/s41398-017-0056-8. PMID 29317604
- [Derived] Mrazek DA, Biernacka JM, McAlpine DE, Benitez J, Karpyak VM, Williams MD, Hall-Flavin DK, Netzel PJ, Passov V, Rohland BM, Shinozaki G, Hoberg AA, Snyder KA, Drews MS, Skime MK, Sagen JA, Schaid DJ, Weinshilboum R, Katzelnick DJ. Treatment outcomes of depression: the pharmacogenomic research network antidepressant medication pharmacogenomic study. J Clin Psychopharmacol. 2014 Jun;34(3):313-7. doi: 10.1097/JCP.0000000000000099. PMID 24743713
- [Derived] Ji Y, Biernacka J, Snyder K, Drews M, Pelleymounter LL, Colby C, Wang L, Mrazek DA, Weinshilboum RM. Catechol O-methyltransferase pharmacogenomics and selective serotonin reuptake inhibitor response. Pharmacogenomics J. 2012 Feb;12(1):78-85. doi: 10.1038/tpj.2010.69. Epub 2010 Sep 28. PMID 20877297